CLINICAL TRIAL: NCT02899702
Title: Effectiveness of Intravenous Immunoglobulins (IVIG) in Toxic Shock Syndromes in Children: a Multicentre European Randomized Controlled Trial
Brief Title: Effectiveness of Intravenous Immunoglobulins (IVIG) in Toxic Shock Syndromes in Children
Acronym: IGHN2
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no EC approval obtained
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL16_0079
Record Dates: First submitted 2016-09-02; First posted 2016-09-14 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Staphylococcal Infection; Streptococcal Infection
MeSH Terms: conditions — Staphylococcal Infections; Streptococcal Infections | interventions — Immunoglobulins, Intravenous; Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVIG (Experimental): PRIVIGEN (CSL Behring) NORMAL HUMAN IMMUNOGLOBULINS L-PROLINE, Water for injection
  Interventions: Drug: PRIVIGEN (CSL Behring)
- control (Placebo Comparator): Single administration of Albumin 4% diluted albumin (LFB), within 12 hours following PICU admission (or outbreak of first shock signs). Isovolume - so dose of 0.8 g/kg We chose as placebo albumin diluted to 4% because this solution has the advantage of having a comparable osmolality.
  The treatment of toxic shock will be standardized. It consists of antibiotics: Amoxicillin-clavulanate and clindamycin (or Rifampicin, Rifadine® if allergic). Antibiotics are not considered as experimental treatments for this study. All treatments essential for the treatment of acute condition will be allowed and are not considered as experimental treatments for this study.
  Interventions: Drug: Albumin

INTERVENTIONS:
Drug: PRIVIGEN (CSL Behring) — Single administration of intravenous immunoglobulin solution Privigen® (CSL Behring AG, Bern, Switzerland) at a dose of 2g / kg. IGIV 2g/kg within 12 hours following PICU admission (or outbreak of first shock signs).
  The treatment of toxic shock will be standardized. It consists of antibiotics: Amoxicillin-clavulanate and clindamycin (or Rifampicin, Rifadine® if allergic). Antibiotics are not considered as experimental treatments for this study. All treatments essential for the treatment of acute condition will be allowed and are not considered as experimental treatments for this study.
  Arms: IVIG
Drug: Albumin — 4%(LFB) ALBUMIN Single administration of human Albumin 4% diluted albumin (VIALEBEX® LFB), within 12 hours following PICU admission (or outbreak of first shock signs). Isovolume - so dose of 0.8 g/kg (4gG, 100 ML, Sodium chloride 0.61 G / 100ML Water for injections QSP 100 ML Sodium caprylate 0.3 G / 100ML) We chose as placebo albumin diluted to 4% because this solution has the advantage of having a comparable osmolality.
  The treatment of toxic shock will be standardized. It consists of antibiotics: Amoxicillin-clavulanate and clindamycin (or Rifampicin, Rifadine® if allergic). Antibiotics are not considered as experimental treatments for this study. All treatments essential for the treatment of acute condition will be allowed and are not considered as experimental treatments for this study.
  Arms: control

SUMMARY:
IGHN2 is an international, multicenter, double blind, randomized controlled trial aimed at assessing the efficacy on organ dysfunctions of Intravenous Immunoglobulins (IVIG) treatment in the acute phase of streptococcal or staphylococcal toxic shock syndrome in children.

ELIGIBILITY:
Inclusion Criteria:

* Child/adolescent: 1 month < Age < 17 year-old,
* admitted to PICU with a strong suspicion of staphylococcal or streptococcal infection; at least one following criterion, with at least one following criteria:

  1. Toxic Shock Syndrom as defined by Centre for Disease Control criteria
  2. or group A Streptococcus necrotizing fasciitis (positive streptest)
  3. or varicella with infected lesions and rash or positive streptest
  4. or erythrodermic rash in menstrual period
  5. or pleuropneumonia with erythrodermic rash or positive streptest in pleural fluid
  6. or erythrodermic rash and biological fluid positive to streptococcus A or staphylococcus (articular, pericardial, bronchopulmonary, pharynx)
* With shock resistant to fluid resuscitation, defined as existence, despite 40 ml/kg of fluid bolus within 1 hour, of:

  1. hypotension (< 5th percentile)
  2. or systolic blood pressure < 2 SD regarding age
  3. or need for vasoactive drugs in order to maintain blood pressure at a normal level (dopamine > 5µg/kg/min or dobutamine, adrenaline, noradrenaline, milrinone whatever the dose)
  4. or 2 signs of hypo perfusion among:

     1. metabolic acidosis with base deficit > 5
     2. lactate x 2 normal laboratory value
     3. diuresis < 0,5 ml/kg/h
     4. capillary refill time > 5 sec
     5. Skin/central temperature difference > 3°C
* With informed consent signed by at least one parent before any procedures or treatments related to the study.

Exclusion Criteria:

* First signs of shock appeared more than 24h ago
* Known hypersensitivity to one of the components (study treatment or placebo , see below)
* Hypersensitivity to homologous immunoglobulins, specifically in very rare cases of Ig A deficit, when the patient has anti-IgA antibodies
* Known hyperprolinemia
* Immunodeficiency (acquired or not),
* Immunosuppressive drugs
* No health cover

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
organ dysfunctions | between day of admission and day 3
  Average variation in Pediatric Logistic Organ Dysfunction 2 ( PELOD-2) score compared between the IVIG treatment arm and the placebo arm.

SECONDARY OUTCOMES:
global mortality | 1 year
disability assessed by the Pediatric Overall Performance Category (POPC) score | one year after recruitment
impairment assessed by the Vineland Adaptive Behavior Scale 2 (VABS II) | one year after recruitment
organ dysfunctions assessed by the PELOD-2 score | over the first 5 days in Paediatric Intensive Care Unit (PICU)

CONTACTS AND LOCATIONS:
Overall Officials: Etienne JAVOUHEY, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No